CLINICAL TRIAL: NCT02091544
Title: Kijk op Overgewicht Bij Kinderen: Study Regarding Etiological Factors, Risk Factors and Early Stages of Chronic Disease in Different Degrees of Childhood Overweight
Brief Title: Etiological Factors, Risk Factors and Early Stages of Chronic Disease in Different Degrees of Childhood Overweight
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: COACH
Record Dates: First submitted 2013-09-17; First posted 2014-03-19 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Childhood Obesity
Keywords: overweight; obesity; children; lifestyle intervention
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Urine
  * Feces
  * Blood&DNA
  * Liver ultrasound & fibroscan
  * Lipidomics
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lifestyle intervention: lifestyle intervention
  Interventions: Other: Lifestyle intervention

INTERVENTIONS:
Other: Lifestyle intervention

SUMMARY:
Children and adolescents with overweight and obesity are predisposed to significant health problems. It is known that childhood obesity can adversely affect almost every organ system, and if left untreated, the major impact of childhood overweight is likely to be felt in the next generation of adults.

The aim of " Kijk op overgewicht bij kinderen" is to collect and follow-up longitudinal data from a population of different degrees of children with overweight regarding etiological factors, risk factors and early stages of chronic disease in different degrees of childhood overweight.

DETAILED DESCRIPTION:
Furthermore, from april 2020 onwards, a prospective sub study will be conducted. This sub study aims to investigate the changes in lifestyle behaviour of children with overweight or obesity and their families during the COVID-19 pandemic, including the (governmental) measures taken for this, and the effect of obesity and different weight-related risk factors on the host response of these children.

The goal of this sub study is to collect data to enable analyses for future research questions regarding the influence of the COVID-19 on the lifestyle of a child with overweight and their family. Endpoints are for example physical activity, eating behavior, BMI-z score, remote lifestyle coaching, quality of life and parental practices regarding nutrition and physical activity behavior. We will also measure symptoms associated with COVID-19 and the host response that target COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the COACH program
* Aged till 18 years old (at time of inclusion)
* Overweight or obesity according to International Obesity Task Force (IOTF) criteria

Exclusion Criteria:

• None

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: overweight or obese children according to the International Obesity Task Force (IOTF) criteria < 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-04; Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
The number of overweight or obese children | approximately 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Anita Vreugdenhil, Dr, Principal Investigator — Maastricht University Medical Center; Luc Zimmermann, Prof.dr., Study Chair — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] van Dam MJCM, Pottel H, Delanaye P, Vreugdenhil ACE. The evaluation of kidney function estimation during lifestyle intervention in children with overweight and obesity. Pediatr Nephrol. 2024 Nov;39(11):3271-3278. doi: 10.1007/s00467-024-06435-0. Epub 2024 Jul 4. PMID 38963556
- [Derived] Lubrecht J, Arayess L, Reijnders D, Hesselink ML, Velde GT, Janse A, von Rosenstiel I, van Mil EGAH, Verweij M, Vreugdenhil ACE. Weight Gain in Children during the COVID-19 Pandemic and the Protective Effect of Lifestyle Intervention in Children with Obesity. Obes Facts. 2022;15(4):600-608. doi: 10.1159/000525298. Epub 2022 May 31. PMID 35640561
- [Derived] van Dam MJCM, Pottel H, Vreugdenhil ACE. Creatinine-based GFR-estimating equations in children with overweight and obesity. Pediatr Nephrol. 2022 Oct;37(10):2393-2403. doi: 10.1007/s00467-021-05396-y. Epub 2022 Feb 24. PMID 35211793
- [Derived] Ten Velde G, Plasqui G, Dorenbos E, Winkens B, Vreugdenhil A. Objectively measured physical activity and sedentary time in children with overweight, obesity and morbid obesity: a cross-sectional analysis. BMC Public Health. 2021 Aug 17;21(1):1558. doi: 10.1186/s12889-021-11555-5. PMID 34404361
- [Derived] Rijks JM, Plat J, Dorenbos E, Penders B, Gerver WM, Vreugdenhil ACE. Association of TSH With Cardiovascular Disease Risk in Overweight and Obese Children During Lifestyle Intervention. J Clin Endocrinol Metab. 2017 Jun 1;102(6):2051-2058. doi: 10.1210/jc.2016-3057. PMID 28379580
- [Derived] Rijks J, Karnebeek K, van Dijk JW, Dorenbos E, Gerver WJ, Stouthart P, Plat J, Vreugdenhil A. Glycaemic Profiles of Children With Overweight and Obesity in Free-living Conditions in Association With Cardiometabolic Risk. Sci Rep. 2016 Aug 18;6:31892. doi: 10.1038/srep31892. PMID 27534260
- [Derived] Rijks J, Penders B, Dorenbos E, Straetemans S, Gerver WJ, Vreugdenhil A. Pituitary response to thyrotropin releasing hormone in children with overweight and obesity. Sci Rep. 2016 Aug 3;6:31032. doi: 10.1038/srep31032. PMID 27485208
- See also: COACH website — http://www.coachmaastricht.com